CLINICAL TRIAL: NCT01495845
Title: Implementation of a Personalized Medicine (Pharmacogenomics) Service in a Community Pharmacy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Kerr Drug (Unknown); Laboratory Corporation of America (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 10-1558
Record Dates: First submitted 2011-12-16; First posted 2011-12-20 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Stroke; Transient Ischemic Attack; Myocardial Infarction
Keywords: pharmacogenomics; feasibility; community pharmacy; personalized medicine; clopidogrel; Plavix
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient; Myocardial Infarction | interventions — Precision Medicine; Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Pharmacogenomics testing for clopidogrel responsiveness — Patients must come to the pharmacy for all visits. At the 1st visit, the patient will provide consent, a complete list of medications, a complete pre-study questionnaire, a copy of their insurance card, and a buccal swab (collected by the pharmacist). The swab will be sent to the testing facility for genotypic testing of CYP2C19. Upon receipt of the results of the results, the pharmacist will propose an intervention to the prescriber based on the patient's indication for clopidogrel and the identification of certain genetic variations atCYP2C19. All patients will be asked to return to the pharmacy for explanation of the results and implementation of any changes approved by the prescriber and to complete a follow-up questionnaire. After the visit to explain the results of testing, the patient's insurance will be billed electronically for a medication therapy management visit; patients without insurance will not be billed. Patients may opt out of billing to insurance at any time.
  Other Names: Personalized medicine; Pharmacogenetics

SUMMARY:
The purpose of this study is to determine the feasibility of pharmacogenomics testing in a community pharmacy using clopidogrel as an example. The investigators hypothesize that this testing is feasible in this setting.

DETAILED DESCRIPTION:
To determine if the study is feasible, we will examine the change in patient perception of pharmacogenomics testing (before and after the study), the percentage of patients interested in this service, the response rate of providers to pharmacist recommendations, the pharmacist time requirement, and reimbursement rate for pharmacist services.

ELIGIBILITY:
Inclusion Criteria:

* Prescribed clopidogrel (Plavix) by their prescriber
* Aged 18 or older
* Currently on clopidogrel therapy for one of the following indicated uses: post-ACS, Recent PCI with stenting, History of TIA or stroke

Exclusion Criteria:

* Are unable to complete study materials (surveys) with or without assistance, including non-English speaking patients
* Are taking clopidogrel for a reason other than stated in inclusion criteria
* Are pregnant or nursing
* Have an allergy to aspirin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of Pharmacogenomics testing in a Community pharmacy | 3 months
  Change in patient perception of testing, reimbursement for pharmacist time, provider acceptance, and amount of pharmacist time required will be measured as part of the provision of this service.

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie Ferreri, PharmD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Kerr Drug, Chapel Hill, North Carolina, United States